CLINICAL TRIAL: NCT01815528
Title: Single -Arm, Multicenter Phase-II Trial for Catumaxomab and Chemotherapy in Patients With Recurrent Ovarian Cancer to Investigate the Feasibility and Clinical Activity of Initial Intraperitoneal Catumaxomab Followed by Chemotherapy Regimes
Brief Title: Feasibility and Clinical Activity of Initial Intraperitoneal Catumaxomab Followed by Chemotherapy in Patients With Recurrent Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: JSehouli (Other)
Responsible Party: Sponsor-Investigator, JSehouli, Prof. Dr. med. Jalid Sehouli, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Cat-Ovar_2011
Record Dates: First submitted 2013-03-14; First posted 2013-03-21 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2015-02

CONDITIONS: Recurrent Epithelial Ovarian Cancer
Keywords: recurrent epithelial ovarian cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — catumaxomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Catumaxomab (Experimental): Catumaxomab treatment followed by an established chemotherapy regimen
  Interventions: Drug: Catumaxomab

INTERVENTIONS:
Drug: Catumaxomab — Catumaxomab dosing comprises the following four intraperitoneal (i.p.) infusions via an i.p.-port or an indwelling catheter:
  1. 10 µg on day 0
  2. 20 µg on day 3
  3. 50 µg on day 7
  4. 150 µg on day 10

SUMMARY:
Single -arm, multicenter phase-II trial for catumaxomab and chemotherapy in patients with recurrent ovarian cancer to investigate the feasibility and clinical activity of initial intraperitoneal catumaxomab followed by chemotherapy regimes.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed epithelial ovarian cancer, primary peritoneal carcinomatosis or fallopian tube cancer
* Recurrent ovarian cancer disease
* Signs for progression either measurable disease according to RECIST or CA 125 increase according the GCIG-criteria or clinical symptoms of tumor progression according to RECIST
* Radiologically and cytologically confirmed malignant ascites possible to puncture
* Life expectancy ≥ 12 weeks
* Age ≥ 18 years
* ECOG performance status at least 1
* No prior operation or, in case of prior operation, the patient must be recovered therefrom. The operation must be performed at least 4 weeks prior to start of study drug
* Capable of understanding the purposes and risks of the study, willing and able to participate in the study, and written informed consent
* Non-childbearing potential or negative pregnancy test

Exclusion Criteria:

* known brain metastases
* Concomitant cancer, chemo- or radiotherapy (except for local radiation therapy for bone marrow metastases)
* Any investigational product within 2 weeks prior to first administration of catumaxomab
* In cases of previous exposure to investigational product, cancer-, chemo-, immune- or radiotherapy (except for local radiation therapy for bone marrow metastasis):

not sufficiently recovered from previous treatment (toxicity present) based on adequate laboratory values and general status according to other in-/exclusion criteria (i.e. this might be less than 1 or 2 weeks after a weekly or bi-weekly scheduled previous therapy regimen)

* Patients must not have been exposed to nitrosoureas or mitomycin C within 6 weeks prior the first infusion of catumaxomab
* Abnormal organ or bone marrow function
* Use of immune-suppressive agents for the past 4 weeks prior to first administration of catumaxomab. For regular use of systemic corticosteroids patients should only be included after stepwise discontinuation to be free of steroids for a minimum of 5 days prior to study entry
* Any known active and chronic infection
* Known HIV infection and / or hepatitis B virus or hepatitis C virus
* Any other concurrent disease or medical conditions that are deemed to interfere with the conduct of the study as judged by the investigator
* Known or suspected hypersensitivity to catumaxomab and its analogues in general or to murine proteins (from rat or mouse)
* Known or suspected hypersensitivity to PLD, topotecan, paclitaxel, gemcitabine or their excipients.
* Patients with congestive heart failure New York Heart Association (NYHA) Class III and IV. Cardiac arrhythmias (except atrioventricular block type I and II, atrial fibrillation/flutter bundle brunch block)or other signs and symptoms of relevant cardiovascular disease
* Body mass index (BMI) < 17 (assessment after ascites drainage)
* Inadequate respiratory function in the opinion of the investigator
* Presence of complete bowel obstruction
* Patients with substance abuse, medical or psychological or social conditions which the investigator believes would preclude compliance with the study requirements.
* Unwilling or unable to follow protocol requirements
* Participation in another clinical study with experimental therapy within 14 days before start of treatment
* Legal incapacity or limited legal capacity
* Subjects housed in an institution on official or legal orders
* Pregnancy or lactation period

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-03; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Feasibility of close sequential combination of catumaxomab and established chemotherapy regimens | Approximately 5 months after start of treatment per patient
  Feasibility of close sequential combination of catumaxomab and established chemotherapy regimens defined by rate of patients with at least 4 chemotherapy cycles following 4 applications of catumaxomab within 20 days as described in the scope of this clinical trial.

SECONDARY OUTCOMES:
Number and severity of adverse events as a measure of safety and tolerability | Approximately 2.5 years after start of study
  Overall safety evaluation, including cytokine related toxicities (safety score catumaxomab
  * number and severity of adverse events
  * number of patients with AEs
  * occurrence of cytokine release related symptoms
  * hospitalization frequency and duration
  * changes in clinically relevant laboratory values (hematology, clinical chemistry, coagulation, and urinalysis)
Percentage of patients who can receive all 4 applications of catumaxomab within 20 days and who are able and committed to receive further mono chemotherapy | Approximately 2.5 years after start of study
  Percentage of patients who can receive all 4 applications of catumaxomab within 20 days and who are able and committed to receive further mono chemotherapy
Percentage of patients who can start chemotherapy after a maximum of 4-7 days after last catumaxomab application | Approximately 2.5 years after start of study
  Percentage of patients who can start chemotherapy after a maximum of 4-7 days after last catumaxomab application
Percentage of patients with no signs of malignant ascites at time of progression or change of therapeutic strategy | Approximately 2.5 years after start of study
  Percentage of patients with no signs of malignant ascites at time of progression or change of therapeutic strategy
Puncture-free interval (defined as paracentesis-free interval after last catumaxomab application/ removal of catheter) | Approximately 2.5 years after start of study
  Puncture-free interval (defined as paracentesis-free interval after last catumaxomab application/ removal of catheter)
Time to progression (TTP) according to RECIST and/or CA-125 response rate | Approximately 2.5 years after start of study
  Time to progression (TTP) according to RECIST and/or CA-125 response rate
Overall response rate (ORR) defined as patients with complete or partial response and duration of response (according to RECIST and/or CA-125 response) | Approximately 2.5 years after start of study
  Overall response rate (ORR) and duration of response (according to RECIST and/or CA-125 response) of second or third or fourth line chemotherapy and compare with historical data
To assess treatment free interval to subsequent therapy (defined as duration of the interval between last chemotherapy application and start of next chemotherapy | Approximately 2.5 years after start of study
  To assess treatment free interval to subsequent therapy (defined as duration of the interval between last chemotherapy application and start of next chemotherapy
To assess PFS according to RECIST and/or CA-125 response rate, OS | Approximately 2.5 years after start of study
  To assess PFS according to RECIST and/or CA-125 response rate, OS
To assess quality of life over time as defined by EORTC-QLQ C 30 and Ovar 28 questionnaire | Approximately 2.5 years after start of study
  To assess quality of life over time as defined by EORTC-QLQ C 30 and Ovar 28 questionnaire
Potential predictive clinical factors for response to catumaxomab | Approximately 2.5 years after start of study
  Analysis of potential predictive clinical factors for response to catumaxomab (e.g. amount of ascites, histology, relative lymphocyte count)

CONTACTS AND LOCATIONS:
Locations (1):
- Charité Campus Virchow-Klinikum, Berlin, Germany